CLINICAL TRIAL: NCT00978445
Title: Use of a Novel Remote Home PT/INR-monitoring Device for Long-Term Anticoagulation Management
Brief Title: Remote Home Prothrombin Time (PT)/International Normalized Ratio (INR) Monitoring and Patient Management System
Acronym: vMetrics-AMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ZIN Technologies, Inc. (Industry)
Collaborators: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Carlos Grodsinsky, Vice President of Technology, ZIN Technologies, Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: vMetrics-AMS-01
Record Dates: First submitted 2009-09-15; First posted 2009-09-17 (Estimated); Results first posted 2013-03-21 (Estimated); Last update posted 2013-03-21 (Estimated); Status verified 2013-03

CONDITIONS: Venous Thromboembolism
Keywords: Systemic embolic events; Thromboembolic Complications with Atrial Fibrillation; Prophylaxis with Atrial Fibrillation; Mechanical Cardiac Valve Replacement
MeSH Terms: conditions — Venous Thromboembolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Home/Standard (Experimental): all participants recieved vMetric protocol at home and in clinical setting, in this ARM the standard protocol was at home first then in clinic INR and interaction with a care giver.
  Interventions: Other: vMetrics protocol
- Standard/Home (Experimental): all participants recieved vMetric protocol at home and in clinical setting, in this ARM the standard protocol was an in clinic INR and interaction with a care giver, then the Home protocol was as described.
  Interventions: Other: vMetrics protocol

INTERVENTIONS:
Other: vMetrics protocol — use vmetrics protocol and device or use standard in clinic monitoring

SUMMARY:
Long-term anticoagulation is indicated in patients for the prophylaxis and/or treatment of the thromboembolic complications associated with atrial fibrillation and/or mechanical cardiac valve replacement, prevention or treatment of venous thromboembolism (deep vein thrombosis and pulmonary embolism), to prevent thromboembolic events post-myocardial infarction, and in patients with systemic embolic events. Currently the only approved oral medication for anticoagulation is warfarin (Coumadin, Bristol-Myers Squibb and generic warfarin. Dosage is controlled by periodic determinations of the prothrombin time (PT)/International Normalized Ratio (INR). Under treatment may lead to venous or arterial thrombotic events or stroke, while over treatment may lead to major bleeding and even death. Patients require frequent INR monitoring to maintain a therapeutic level of anticoagulation. The therapeutic INR range varies by clinical indication, most commonly an INR 2-3 goal, but ranging from 1.5-4.0. Bleeding complications are more likely to occur above an INR value of 4.0. The vMetrics - Anticoagulation Management System is a remote patient management solution for Oral Anticoagulation Care patients. This system provides confirmation of patient question and testing protocols as well as virtual patient management care capability for dosage and patient scheduling. This trial will provide end points to ascertain efficiency against standard care protocol and confirm equivalent care standards.

DETAILED DESCRIPTION:
The creation of optimal devices for patient self-testing protocols for anticoagulation management is an area of active medical research. The current pilot study represents the initial step in the development of a new customized device for this purpose, the vMetrics - Anticoagulation Monitoring System. The v-Metrics Anticoagulation Monitoring System (vMetrics AMS) is defined by: 1. A PT/INR home monitoring unit which interfaces to FDA approved PT/INR home monitors such as the Hemosense INRatio device, and 2. an anticoagulation clinic patient management application which manages patient communications, database of prior test results, testing schedules, and communication to an EMR.

The INR home-monitoring system to be tested in this study will address several of the limitations of currently available technologies and practices for standard and home INR self-testing. The proposed project will develop a self-testing device that maximizes safety and efficiency for both the patient and the health care provider. The monitoring device (vMetrics) allows the wireless transmission of the INR result from an approved home INR measuring monitoring device (ex:HemoSense - INRatio) to a secure database in a health care provider staffed anticoagulation clinic. The device will also collect yes/no responses to a set of standard questions from the subject to assure patient safety and determine optimal Coumadin dosing. Upon receipt of the patient data, the Coumadin provider can review the INR result and responses to the questions and use standard Coumadin dosing protocols and clinical judgment to transmit dosing instructions back to the patient through the device. A calendar schedule of dosing until the next scheduled INR check will be transmitted to the patient. In certain instances (i.e., high INR > 5), the device will transmit instructions to call the Coumadin clinic. The subject will confirm receipt of the Coumadin dose sent to him/her by pressing a button on the device (which transmits the confirmation back to the database). This process may reduce inconvenience to the subject, the INR value is reported directly from the device reducing the possibility of error, two-way communication is wireless and will reduce the need for telephone contact, thus potentially saving health care provider and patient time. In addition, the data from the encounter will be available in a form that can be entered into the patient's electronic medical record. The patient will enter data into the device using a 4-digit passcode that will allow for security of data.

In addition to coordinating INR transmission through the home INR device, a customized database will provide a platform for the anticoagulation clinic patient management application (Wireless Home Coumadin clinic). This platform which will organize the workflow of the Coumadin provider to more easily determine which patients are due (or overdue) for monitoring, and which patients have transmitted an INR value and questionnaire and are awaiting a response.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-80 years
* Requires long-term oral anticoagulation therapy for one of the following indications:

  * Venous thromboembolism (deep vein thrombosis or pulmonary embolism)
  * Arterial thromboembolic event(s)
  * Atrial fibrillation
  * Mechanical heart valve
* INR goal set at 2-3 by supervising physician
* Subject has been followed in the Vascular Medicine Coumadin program for at least 3 months
* No INR values > 7, and no major thrombotic or bleeding complications within the preceding 3 months of follow-up in the Coumadin program.
* Subject has been compliant with INR monitoring during period of enrollment in the Vascular Medicine Coumadin program.
* Physically able and willing to perform finger stick INR measurements on self
* Able to use the hand-held monitoring device and have adequate vision to read information on the device screen

Exclusion Criteria:

* Inability to speak and read English
* Anticipated interruption in anticoagulation within the next 6 months (e.g., for elective major surgery, pregnancy)
* Cognitive impairment which makes ability to perform necessary procedures related to the remote home monitoring device unlikely

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2009-09; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heather Gornik, M.D., Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic main campus, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Inrolled 25 patients in two arms of 12 weeks from patient population of Cleveland Clinic Foundation
Pre-assignment Details: Clear enrollement criteria were created only real exclusion was if physician did not believe patient could perform protocol and if outside of age criteria.
Groups:
- Home/Standard: all participants recieved home and standard protocol, in this ARM the home protocol was a virtual INR and communication using a remote communication device called vMetrics.
- Standard/Home: all participants recieved home and standard protocol, in this ARM the standard protocol was a in clinic INR and interaction with a care giver, then the Home protocol was as described.
Period: Overall Study
Arm/Group | Home/Standard | Standard/Home
Started | 12 | 13
Completed | 10 | 12
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- All Participants: all participants recieved all interventions during study
Arm/Group | All Participants
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 53.7 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 15
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Time Spent Per PT/INR Monitoring Encounter
Description: minutes spent measuring coagulation time of blood on standard versus home protocol
Time Frame: Once per week during 12 week study
Population: through minimum power study
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- All Participants-Home Protocol: all participants recieved all interventions during study
- All Particpants - Standard Protocol: First and second group with vMetrics
Arm/Group | All Participants-Home Protocol | All Particpants - Standard Protocol
Number analyzed (Participants) | 22 | 22
minutes | 19.4 (2.3) | 47 (2.6)

2. Secondary Outcome: Change in Quality of Life - Based on Quality of Life Scores PSQ-18 (Short Form Patient Satisfaction Questionnaire) Duke Anticoagulation Satisfaction Scale SF-12 (Short Form 12 Version 2) Quality of Life Questionnaire
Description: we are interested in the relative measure of quality of life by comparing quality of life measures through use of PSQ-18 and other measures listed.
  Higher scores indicate a better quality of life.
Time Frame: During study vist number 2 after 12 week study period, repeated after second study 12 week period study visit #3
Population: power analysis
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- All Participants - Standard Protocol: all participants recieved all interventions during study
Arm/Group | All Participants-home Protocol | All Participants - Standard Protocol
Number analyzed (Participants) | 22 | 22
scores on a scale
  PSQ-18 | 51.1 (.7) | 50.8 (.6)
  DASS | 47.5 (2.6) | 49.7 (2.7)

ADVERSE EVENTS:
Time Frame: During study period - 12 weeks
Description: no adverse events
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No